CLINICAL TRIAL: NCT02492230
Title: Left Atrial Appendage Closure Compared to Standard Antiplatelet Therapy in Patients With AF Who Underwent Percutaneous Coronary Intervention
Brief Title: Left Atrial Appendage Closure Compared to Standard Antiplatelet Therapy in Patients With AF Who Underwent PCI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 241592LLAPCI
Record Dates: First submitted 2015-06-30; First posted 2015-07-08 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): After successful PCI the control group will take Triple therapy (warfarin + clopidogrel+aspirin) during 45 days and after combination of warfarin+clopidogrel to 6 months after procedure and then only warfarin. Patients will be followed at 45 day, and every 3 months during 12 months of follow up.
  Interventions: Drug: Warfarin
- Study Group (Experimental): Left Atrial Appendage Closure Device will be implanted immediately after successful PCI procedure. It will be implanted via a trans-septal approach by use of a catheter based delivery system to seal the ostium of the LAA. The implantation will be guided by fluoroscopy and TEE to verify proper positioning and stability. The study group will take Triple therapy (warfarin+clopidogrel+aspirin) during 45 days following PCI and after control TEE, warfarin will be discontinued. Then patients from the study group will take DAPT combination (clopidogrel+aspirin) to 6 months after procedure and then only aspirin. Patients will be followed at 45 day, and every 3 months during 12 months of follow up
  Interventions: Device: Left Atrial Appendage Closure Device (Watchman)

INTERVENTIONS:
Device: Left Atrial Appendage Closure Device (Watchman) — This device is a self-expanding nickel titanium (nitinol) frame structure with fixation barbs and a permeable polyester fabric cover. The device ranges in diameter from 21 mm to 33 mm to accommodate varying LAA anatomy and size. It will be implanted via a trans-septal approach by use of a catheter based delivery system to seal the ostium of the LAA. The implantation will be guided by fluoroscopy and TEE to verify proper positioning and stability. The dose of warfarin will be adjusted to maintain INR 2.0 - 3.0 for 45 days. If TEE data shows no additional flow in LAA, warfarin will be discontinued: Aspirin dose: 75 mg for all period of study; Clopidogrel dose: 75 mg for 6 months after procedure.
  Other Names: PCI
  Arms: Study Group
Drug: Warfarin — Warfarin dose adjusted to maintain INR 2.0-3.0 for all period of study; Aspirin dose-75mg for 45 days after randomization; Clopidogrel dose-75mg for 6 months after procedure.
  All drugs will be started before PCI procedure. Low molecular weight heparins will be used before procedure and will be stopped when INR reach 1.8-2.0.
  Other Names: PCI
  Arms: Control Group

SUMMARY:
The objective of Left atrial appendage closure compared to standard antiplatelet therapy in patients with AF who underwent percutaneous coronary intervention (LLA-PCI) study is to evaluate the safety and efficacy of implantation of left atrial appendage closure compared to standard antiplatelet therapy for prevention of thromboembolic events and stent thrombosis in subjects with AF who underwent PCI.

DETAILED DESCRIPTION:
This will be prospective randomized (1:1) open label pilot study. Patients with unstable angina and non-ST-elevation ACS and history of AF will be included in this study. After PCI and DES implantation TEE will be performed for assessing LAA anatomy and size eligible for left atrial appendage closure device implantation. After screening all patients will be randomized in two groups. The first (control) group will receive standard antiplatelet and anticoagulation therapy according to the guidelines (2), the second group of patients will undergo left atrial appendage closure device implantation. After the PCI the first group will take Triple therapy (warfarin + clopidogrel+aspirin) during 45 days and after combination of warfarin+clopidogrel to 6 months after procedure and then only warfarin. The second group will take Triple therapy (warfarin+clopidogrel+aspirin) during 45 days following PCI and after control TEE, warfarin will be discontinued. Then patients from the second group will take DAPT combination (clopidogrel+aspirin) to 6 months after procedure and then only aspirin. Patients will be followed at 45 day, and every 3 months during 12 months of follow up (Figure 1). At each follow-up visits the data regarding clinical events and healthcare utilization will be collected.

ELIGIBILITY:
Inclusion criteria:

* age > 18 years old
* Acute coronary syndrome without ST elevation and unstable angina 2 weeks before enrolment
* Successful PCI procedure with DES
* History of atrial fibrillation (paroxysmal, persistent or permanent) with ECG documentation within previous 12 month
* CHA2DS2-VASC ≥ 2
* HAS-BLED ≥ 3
* LAA eligible for left atrial appendage closure device implantation (TEE data)

Exclusion criteria:

* age <18 or >80 years old
* INR >3
* recurrent myocardial infarction
* myocardial infarction with ST elevation
* EF<50%
* severe comorbidities
* Cardiogenic shock (within 72 hours of randomization), as defined by the need for intraaortic balloon support or the requirement for intravenous inotropic support.
* anemia < 100 g/l
* uncontrolled hypertension
* thrombocytopenia
* oncology
* obesity, BMI>40
* LAA thrombosis
* Women of childbearing potential (unless post-menopausal or surgically sterile)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with bleeding according TIMI and GUSTO scales | 12 months

SECONDARY OUTCOMES:
Cardiovascular death | 12 month
Sudden cardiac death | 12 month
Death due to heart failure | 12 month
Death due to stroke | 12 month
Death due to cardiovascular procedures | 12 month
Death due to CV hemorrhage | 12 month
Death due to other CV causes | 12 month
Periprocedural complications on first FU visit | 1,5 month
All neurologic events with documented diagnosis of stroke or transient ischemic attack | 12 month
Definite stent thrombosis | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Pokushalov, MD, PhD, Study Director — State Research Institute of Circulation Pathology
Locations (1):
- State Research Institute of CIrculation Pathology Novosibirsk, Russian Federation, Novosibirsk, Russia